CLINICAL TRIAL: NCT03805685
Title: The Influence of Preoperative Risk Factors on Perioperative Neurocognitive Disorders in Patients Scheduled for Non-cardiac Surgery
Brief Title: Preoperative Risk Factors and Perioperative Neurocognitive Disorders
Status: Completed | Type: Observational
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: CHU de Charleroi (Other)
Responsible Party: Principal Investigator, Sarah Saxena, Anesthesiologist; Principal Investigator, Université Libre de Bruxelles
Other Study IDs: Lifestyle-Delirium
Record Dates: First submitted 2019-01-05; First posted 2019-01-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Change

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample (as usual)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Non-Cardiac Surgery — Non-cardiac surgery

SUMMARY:
Perioperative neurocognitive disorders (PND's) remain an important complication after surgery. After many years of speculating about the etiology of this complication, currently studies are pointing to an inflammatory cascade being set in motion.

This prospective study is designed to examine preoperative lifestyle factors (such as sedentary behavior) associated with postoperative cognitive impairment in a group of patients undergoing non-cardiac surgery.

The objectives in our study are to:

identify perioperative risk factors for the development of PND's measure the incidence and duration of perioperative neurocognitive disorders in a known high-risk group of elective surgical patients measure a peripheral inflammatory marker (interleukin 6: IL-6) in the same group of surgical patients

DETAILED DESCRIPTION:
Perioperative neurocognitive disorders remain an important complication after surgery. After many years of speculating about the etiology of this complication, currently studies are pointing to an inflammatory cascade being set in motion. Following the combination of surgery/ anesthesia, high molecular group box protein 1 (HMGB1) is released. This damage-associated molecular pattern (DAMP) binds to pattern recognition receptors (PRR) on circulating bone marrow-derived monocytes (BM-DMs). Through an intracellular signaling pathway, the transcription factor NF-kappaB passes into the nucleus, is activated and increases expression and release of pro-inflammatory cytokines. These in turn disrupt the blood brain barrier. Within the brain parenchyma the chemokine MCP-1 (also referred to as CCL2) is upregulated and attracts the BM-DMs through binding to its receptor, CCR2. In turn, this activates the resident quiescent microglia. Together, the BM-DMs and activated microglia release HMGB1 and pro-inflammatory cytokines that disrupt long-term potentiation (LTP) thereby blocking synaptic plasticity changes that are required for the cognitive functions of learning and memory.

Unfortunately, treatment currently is lacking, however optimising lifestyle seems to be a promising pathway in a murine population.

This prospective study is designed to examine preoperative lifestyle factors (such as sedentary behavior) associated with postoperative cognitive impairment in a group of patients undergoing non-cardiac surgery.

Prior to surgery, patients will have a baseline MMSE (mini mental state examination) assessment. At the same time, a standardized history form will be completed to document pertinent patient information, with special emphasis on patterns of smoking and ethanol consumption. French IPAQ data will be collected as well as the Geriatric Depression Scale.

Right before the surgery, a peripheral blood sample will be drawn (to analyse IL-6 levels).

Induction and Maintenance of General Anesthesia: All patients will receive general anesthesia using an endotracheal tube to facilitate ventilatory support.

Induction of anesthesia will be performed using the following:

I.V. (intravenous) Sufentanil 0.1- 0.2 mcg/kg I.V. Lidocaine 1.5 mg/kg I.V. Propofol 2-3 mg/kg I.V. Rocuronium 0.6 -1.2 mg/kg General anesthesia will be maintained using 0.5-2.5% sevoflurane in an O2:air mixture, the latter titrated to maintain an oxygen saturation (SpO2) value of 96% or greater via pulse oximetry.

Additional analgesia will be provided with I.V. Acetaminophen 15 mg/kg and I.V. Diclofenac 1 mg/kg and, if necessary, I.V. sufentanil 5 mcg.

Non-invasive blood pressure will be measured on the upper arm, and a phenylephrine infusion of 0-100 mcg/min will be administered to maintain mean arterial blood pressure within 20% of the preoperative value.

If muscle relaxation is required by the surgeon, I.V. rocuronium may be administered in 10-20 mg boluses. I.V. Sugammadex 4 mg/kg will be administered if needed to reverse neuromuscular blockade.

At the end of the surgery, just prior to emergence from general anesthesia, each patient will receive I.V. ondansetron 4 mg for anti-emetic purposes.

Upon emergence from anesthesia, all patients will be transferred to the post-operative recovery unit.

Depth of anesthesia monitoring will be done via BIS monitor. The BIS monitor value will be maintained in the range of 40-60 to ensure uniform sedation levels in all subjects.

Monitoring of Other Physiological Parameters During General Anesthesia: Heart rate, oxygen saturation (SpO2), respiratory rate, non-invasive blood pressure, end-tidal CO2 levels, inspired/end-tidal O2 levels, inspired/end-tidal sevoflurane concentrations, temperature, and BIS values will be continuously monitored and recorded throughout the surgical procedure, to ensure that the measured physiological parameters are within the normal range. Similarly, the cumulative doses of all sedative and analgesic medications will also be recorded.

Six hours post-operatively, a peripheral blood sample will be drawn again (to analyse IL-6 levels) as well as 24 hours post-operatively.

Once discharged from the hospital, patients will come for a follow-up visit at six weeks post-operatively as well as three months. During this follow-up visit, patients will repeat MMSE testing.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent
* Patients scheduled for non-cardiac surgery (with a duration of 1 to 4 hours)

Exclusion Criteria:

* Lack of comprehension of the French, English or Dutch language
* Visual or auditory impairment
* Any other reason that makes patients unable to perform cognitive testing

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients participating in the study will have to provide written informed consent. Patients of both genders aged 55 or more scheduled for non-cardiac surgery between 8 and 10 AM (with a duration of 1 to 4 hours) will be eligible for enrolment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-02-03 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Pre-operative MMSE | 12 hours
  Mini mental state examination will be evaluated prior to the surgery
MMSE 6 weeks post-operative | 6 weeks
  Mini mental state examination will be evaluated 6 weeks after surgery
MMSE 3 months post-operative | 3 months
  Mini mental state examination will be evaluated 3 months after surgery

SECONDARY OUTCOMES:
Concentration of patient's baseline pre-operative peripheral IL-6 | 12 hours
  Blood samples to measure IL-6 will be drawn prior to the surgery
Concentration of patient's post-operative peripheral IL-6; 6 hours post-operative | 24 hours
  Blood samples to measure IL-6 will be drawn 6 hours after the surgery
Concentration of patient's post-operative peripheral IL-6 ; 24 hours post-operative | 24 hours
  Blood samples to measure IL-6 will be drawn 24 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean Boogaerts, MD; PhD, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- CHU-Charleroi Hopital Civil Marie Curie, Charleroi, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saxena S, Rodts C, Nuyens V, Lazaron J, Sosnowski V, Verdonk F, Seidel L, Albert A, Boogaerts J, Kruys V, Maze M, Vamecq J. Preoperative sedentary behavior is neither a risk factor for perioperative neurocognitive disorders nor associated with an increase in peripheral inflammation, a prospective observational cohort study. BMC Anesthesiol. 2020 Nov 14;20(1):284. doi: 10.1186/s12871-020-01200-w. PMID 33187477